CLINICAL TRIAL: NCT04335903
Title: The Turkish Version of the Vividness of Visual Imagery Questionnaire-2
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 52025
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Body Image; Assessment, Self
Keywords: Imagination; Motor imagery; Body Image; Kinesthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Vividness of Visual Imagery Questionnaire-2 (VMIQ-2) is originally developed in English to determine the vividness of visual imagery. The purpose of this study is to translate and cross-culturally adapt the VMIQ instrument into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The Vividness of Visual Imagery Questionnaire-2 (VMIQ-2) was originally developed in English to determine the vividness of visual imagery. The purpose of this study is to translate and cross-culturally adapt the VMIQ-2 instrument into Turkish and investigate its psychometric properties. One hundred fifty healthy participants will be included. For cross-cultural adaptation, two bi-lingual translators will use the back-translation procedure. Within a 5-to-7-day period after the first assessment, the participants will complete the Turkish version of VMIQ (VMIQ-2-T) to evaluate test-retest reliability. Cronbach's alpha (α) will use to assess internal consistency. The correlation with the Turkish version of Kinesthetic and Visual Imagery Questionnaire-20 will be determined to check the validity.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old
* ability to read and write in Turkish
* no pathology in visual ability and hearing
* able to follow simple instructions

Exclusion Criteria:

* having a chronic disease
* severe musculoskeletal, neurological or cardiovascular disorders that limit mobility
* having any cognitive problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will consist of volunteer, healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2021-08-21 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
The Vividness of Visual Imagery Questionnaire-2 | Baseline (First assessment)
  This questionnaire is composed of 12 items - walking, running, kicking a stone, bending down to pick up a coin, running up stairs, jumping sideways, throwing a stone into water, kicking a ball in the air, running downhill, riding a bike, swinging on a rope, and jumping off a high wall. It requires individuals to imagine themselves performing the 12 items, from three imagery perspectives: internal visual imagery (a first-person perspective), external visual imagery (a third-person perspective), and kinesthetic imagery (feeling the movement).

SECONDARY OUTCOMES:
The Vividness of Visual Imagery Questionnaire-2 | Within a 5-to-7-day period after the first assessment (Second assessment)
  This questionnaire is composed of 12 items - walking, running, kicking a stone, bending down to pick up a coin, running up stairs, jumping sideways, throwing a stone into water, kicking a ball in the air, running downhill, riding a bike, swinging on a rope, and jumping off a high wall. It requires individuals to imagine themselves performing the 12 items, from three imagery perspectives: internal visual imagery (a first-person perspective), external visual imagery (a third-person perspective), and kinesthetic imagery (feeling the movement).
The Movement Imagery Questionnaire-3 | Baseline (First assessment)
  This questionnaire is composed of 4 items and requires individuals to imagine themselves performing the 4 items, from three imagery perspectives: internal visual imagery (a first-person perspective), external visual imagery (a third-person perspective), and kinesthetic imagery (feeling the movement).

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No